CLINICAL TRIAL: NCT02343406
Title: INTELLANCE-2: ABT-414 Alone or ABT-414 Plus Temozolomide Versus Lomustine or Temozolomide for Recurrent Glioblastoma: A Randomized Phase 2 Study of the EORTC Brain Tumor Group
Brief Title: Adult Study: ABT-414 Alone or ABT-414 Plus Temozolomide vs. Lomustine or Temozolomide for Recurrent Glioblastoma Pediatric Study: Evaluation of ABT-414 in Children With High Grade Gliomas
Acronym: INTELLANCE-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-483; 2014-004438-24 (EudraCT Number); EORTC 1410-BTG (Other Grant/Funding Number: European Organization for Research and Treatment of Cancer)
Record Dates: First submitted 2014-12-22; First posted 2015-01-22 (Estimated); Results first posted 2020-05-22 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Epithelial Growth Factor vIII mutation; Temozolomide; Lomustine; ABT-414; European Organization for Research and Treatment of Cancer; Recurrent glioblastoma; Epithelial Growth Factor; Brain Tumor; Brain Tumor Group; Antibody Drug Conjugate; EORTC; Pediatric High Grade Gliomas; Pediatric Diffuse Intrinsic Pontine Glioma; Pediatric WHO grade III glioma; Pediatric WHO grade IV glioma; EGFR amplification; Children
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — depatuxizumab mafodotin; ABT-414; Temozolomide; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- ABT-414/temozolomide (Experimental): Depatuxizumab mafodotin (ABT-414) administered once every 2 weeks in combination with temozolomide (TMZ) to adult participants
  Interventions: Drug: Depatuxizumab mafodotin; Drug: Temozolomide
- ABT-414_adult (Experimental): Depatuxizumab mafodotin (ABT-414) administered once every 2 weeks to adult participants
  Interventions: Drug: Depatuxizumab mafodotin
- Control_lomustine (Active Comparator): Adult participants relapsing during temozolomide (TMZ) treatment or within the first 16 weeks after the first day of the last TMZ cycle received lomustine on Day 1 of every 42-day treatment period until one of the treatment withdrawal criteria was met, up to a maximum of 1 year.
  Interventions: Drug: Lomustine
- Control_ temozolomide (Active Comparator): Adult participants relapsing 16 weeks or more after the first day of the last temozolomide (TMZ) cycle received TMZ on Day 1 to Day 5 for the first 28-day cycle, with dose escalation in subsequent cycles in case of adequate tolerance and treatment continuing until one of the treatment withdrawal criteria was met.
  Interventions: Drug: Temozolomide
- ABT-414_ pediatric (Experimental): Depatuxizumab mafodotin (ABT-414) administered once every 2 weeks to pediatric participants. Temozolomide (TMZ) was only allowed for pediatric participants if its use was in accordance with local clinical practice, and was not considered an investigational product for the study (unless this was a local requirement).
  Interventions: Drug: Depatuxizumab mafodotin

INTERVENTIONS:
Drug: Depatuxizumab mafodotin — Adults: intravenous administration (1.25 mg/kg or 1.0 mg/kg body weight) over 30 to 40 minutes once every 2 weeks until one of the treatment withdrawal criteria was met. The dose was 1.25 mg/kg in the original protocol (Version 1) and Version 2, Amendment 1, and was lowered to 1.0 mg/kg in protocol Version 3, Amendment 2. Pediatric participants: Intravenous administration (1.0 mg/kg body weight for those who were 6 to 17 years old at the date of first dose, or 1.3 mg/kg for those who were 0 to 5 years old) over 30 to 40 minutes or as directed by the guidelines once every 2 weeks until one of the treatment withdrawal criteria was met, for a maximum of one year. If used in combination with temozolomide, depatuxizumab mafodotin was dosed on Day 1 and Day 15 of the TMZ cycle (assuming a standard regimen of 200 mg/m^2/day for 5 days of each 28-day cycle; for other TMZ schedules, timing of the depatuxizumab mafodotin dosing schedule were to be discussed with the medical monitor).
  Other Names: ABT-414
  Arms: ABT-414/temozolomide; ABT-414_ pediatric; ABT-414_adult
Drug: Temozolomide — Capsules administered orally, 150 mg/m^2 on Days 1-5 for the first 28-day cycle, with dose escalation to 200 mg/m^2 in subsequent cycles in case of adequate tolerance until one of the treatment withdrawal criteria was met.
  Other Names: TMZ
  Arms: ABT-414/temozolomide; Control_ temozolomide
Drug: Lomustine — Capsules administered orally, 110 mg/m^2 on Day 1 of every 42-day treatment period. Treatment continued until one of the treatment withdrawal criteria was met, for a maximum of one year.
  Other Names: Gleostine
  Arms: Control_lomustine

SUMMARY:
This study was conducted to evaluate the efficacy and safety of depatuxizumab mafodotin (ABT-414) alone or with temozolomide versus temozolomide or lomustine alone in adult participants with recurrent glioblastoma. The study also included a substudy to evaluate safety, tolerability and pharmacokinetics of ABT-414 in a pediatric population.

DETAILED DESCRIPTION:
The study objectives were to assess whether depatuxizumab mafodotin (ABT-414) alone or in combination with temozolomide (TMZ) improved overall survival (OS), progression-free survival (PFS), tumor response, quality of life, neurological deterioration-free survival (NDFS), and steroid use compared to standard treatment with lomustine single agent or TMZ re-challenge in adult subjects ≥ 18 years of age with centrally-confirmed recurrent epidermal growth factor receptor (EGFR)-amplified glioblastoma. The safety, pharmacokinetics, and efficacy of depatuxizumab mafodotin in children <18 years of age was evaluated in a pediatric substudy. The EMEA-001732-PIP02-15 pediatric investigation plan was withdrawn on 07 July 2019 due to the discontinuation of the depatuxizumab mafodotin research program.

ELIGIBILITY:
Inclusion Criteria:

Adult participants (greater than or equal to 18 years old):

* Histologically confirmed de novo (primary) glioblastoma with unequivocal tumor progression or recurrence.
* In case of testing at the time of first progression: either at least 3 months after the end of radiotherapy or have tumor progression that is clearly outside the radiation field or have tumor progression unequivocally proven by surgery/biopsy
* Absence of any psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule; such conditions should be assessed with the patient before registration in the trial.
* Availability of adequate biological material (formalin-fixed paraffin embedded [FFPE] tumor) for central testing of Epithelial Growth Factor Receptor (EGFR) amplification
* Presence of EGFR amplification confirmed by central assessment; participants with undetermined EGFR status are excluded
* World Health Organization (WHO) Performance status 0 - 2
* No more than one line of chemotherapy (concurrent and adjuvant Temozolomide based chemotherapy including in combination with another investigational agent is considered one line of chemotherapy). Chemotherapy must have been completed at least 4 weeks prior to randomization.
* Post surgery MRI within 48 hours following surgery, however an MRI scan has to be done within 2 weeks prior to randomization.
* Surgery completed at least 2 weeks before randomization and patients should have fully recovered as assessed by investigators.
* Renal function: calculated creatinine clearance ≥ 30 mL/min by the Cockcroft-Gault formula.
* Liver function: bilirubin < 1.5× upper limit of the normal range (ULN), alkaline phosphatase and transaminases (ASAT) < 2.5× ULN

Pediatric sub-study participants (less than 18 years old):

* Histologically proven high grade glioma (HGG: WHO grade III glioma [e.g anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma], grade IV glioma [e.g. glioblastoma, gliosarcoma] or diffuse intrinsic pontine glioma [DIPG]).
* Must either have recurrent/progressive tumor or, if newly diagnosed, have completed any planned radiation therapy at least 4 weeks prior to first dose of ABT-414.
* The tumor tissue must have been determined to have EGFR amplification, (by local or other testing service).
* Availability of adequate biological material for retrospective confirmatory central testing of EGFR amplification
* Participant has sufficiently recovered from previous therapy. The investigator believes that benefit of treating the pediatric subject with ABT-414 outweighs the expected risks and that this treatment is in the best interests of the pediatric subject.
* Renal function: calculated creatinine clearance ≥ 30 mL/min by the Cockcroft-Gault formula for pediatric patients ≥12 years of age and estimated glomerular filtration rate ≥ 30 mL/min/1.73 m^2 by modified Schwartz equation for pediatric patients < 12 years of age.
* Liver function: Total bilirubin ≤ 1.5× upper limit of the normal range (ULN), Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) <= 3× ULN. Participants with Gilbert's syndrome documented in medical history may be enrolled if total bilirubin is < 3 times ULN. Not allowed are participants with known chronic liver disease and/or cirrhosis.

Exclusion Criteria:

Adult population (greater than or equal to 18 years old):

* Prior treatment with nitrosoureas
* Prior treatment with bevacizumab
* Previous exposure to Epithelial Growth Factor Receptor (EGFR) targeted agents, including EGFRvIII targeting agents
* Prior discontinuation of temozolomide chemotherapy for toxicity reasons
* Prior Radiation Therapy (RT) with a dose over 65 Gy to the brain, stereotactic radiosurgery or brachytherapy unless the recurrence is histologically proven
* Previous other malignancies, except for any previous malignancy which was treated with curative intent more than 5 years prior to randomization, and except for adequately controlled limited basal cell carcinoma of the skin, squamous carcinoma of the skin or carcinoma in situ of the cervix
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to randomization.
* No history of wheat allergies and Coeliac disease.
* No EIAED, patients who require anti-convulsant therapy must be taking non-enzyme inducing antiepileptic drugs (non-EIAED). Patients previously on EIAED must be fully switched to non-EIAED at least 2 weeks prior to randomization.

Pediatric sub-study (less than 18 years old):

* (For recurrent disease) No prior RT with a dose over 65 Gy to the brain, stereotactic radiosurgery or brachytherapy unless the recurrence is histologically proven
* No current or recent (within 4 weeks or 5 half-lives [whichever is shorter] before enrollment) treatment with another investigational drug
* Female participants of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to randomization.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (102):
- United States (13):
  - Lucile Packard Children's Hosp /ID# 153678, Palo Alto, California
  - Children's Hospital Colorado /ID# 153677, Aurora, Colorado
  - Univ of Colorado Cancer Center /ID# 134882, Aurora, Colorado
  - Sarah Cannon Research Institute at HealthONE - Denver /ID# 141798, Denver, Colorado
  - Rush University Medical Center /ID# 137542, Chicago, Illinois
  - Dana-Farber Cancer Institute /ID# 154210, Boston, Massachusetts
  - Long Island Brain Tumor Center /ID# 134496, Lake Success, New York
  - Weill Cornell Medicine /ID# 152656, New York, New York
  - Cleveland Clinic Main Campus /ID# 137540, Cleveland, Ohio
  - University of Pittsburgh MC /ID# 134491, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC /ID# 134492, Nashville, Tennessee
  - UT Southwestern Medical Center /ID# 136718, Dallas, Texas
  - Swedish Medical Center /ID# 136719, Seattle, Washington
- Australia (10):
  - Port Macquarie Base Hospital /ID# 134569, Port Macquarie, New South Wales
  - Sydney Children's Hospital /ID# 153533, Randwick, New South Wales
  - Royal North Shore Hospital /ID# 147092, Saint Leonards, New South Wales
  - Calvary Mater Newcastle /ID# 134570, Waratah, New South Wales
  - Southern Medical Day Care Ctr /ID# 134495, Wollongong, New South Wales
  - Royal Brisbane and Women's Hospital /ID# 147091, Herston, Queensland
  - Royal Adelaide Hospital /ID# 135208, Adelaide, South Australia
  - Royal Hobart Hospital /ID# 135209, Hobart, Tasmania
  - Barwon Health University Hospital Geelong /ID# 134493, Geelong, Victoria
  - Royal Children's Hospital /ID# 157624, Melbourne, Victoria
- Austria (3):
  - University Hospital St. Polten /ID# 139070, Sankt Pölten, Lower Austria
  - LKH-Univ. Klinikum Graz /ID# 139071, Graz
  - Kepler Universitätsklinikum GmbH - Neuromed Campus /ID# 139068, Linz
- Belgium (6):
  - Cliniques Universitaires Saint Luc /ID# 139391, Woluwe-Saint-Lambert, Brussels Capital
  - Grand Hôpital de Charleroi /ID# 139342, Charleroi, Hainaut
  - UZ Gent /ID# 152944, Ghent, Oost-Vlaanderen
  - AZ St-Jan Brugge-Oostende AV /ID# 137927, Bruges, West-Vlaanderen
  - ZNA Middelheim /ID# 137926, Antwerp
  - UZ Leuven /ID# 137925, Leuven
- Montreal Neurological Institut /ID# 136309, Montreal, Quebec, Canada
- Czechia (4):
  - Fakultni Nemocnice v Motole /ID# 139509, Prague, Praha 5
  - Masarykuv onkologikcy ustav /ID# 139508, Brno
  - FN Hradec Kralove /ID# 139510, Hradec Králové
  - Univ Hosp Ostrava-Poruba /ID# 139507, Ostrava
- Finland (3):
  - Helsinki Univ Central Hospital /ID# 140078, Helsinki
  - Helsinki Univ Central Hospital /ID# 153069, Helsinki
  - Turku University Hospital /ID# 140861, Turku
- France (11):
  - Centre Oscar Lambret /ID# 169619, Lille, Hauts-de-France
  - CHRU Lille - Hôpital Claude Huriez /ID# 137916, Lille, Hauts-de-France
  - Institut de Cancer de l'Ouest /ID# 137914, Saint-Herblain, Loire-Atlantique
  - Hopital de la Timone /ID# 137911, Marseille, Provence-Alpes-Côte d'Azur Region
  - CHU de Nice /ID# 137917, Nice, Provence-Alpes-Côte d'Azur Region
  - Centre Leon Berard /ID# 137918, Lyon, Rhone
  - Institut de Cancer de l'Ouest /ID# 137909, Angers
  - Hospices Civils de Lyon /ID# 137913, Bron
  - Hopital Pitie Salpetriere /ID# 145887, Paris
  - CHU-Hopital Avicenne /ID# 137910, Bobigny, Île-de-France Region
  - Gustave Roussy /ID# 137912, Villejuif, Île-de-France Region
- Germany (5):
  - Universitaetsklinik Heidelberg /ID# 137924, Heidelberg, Baden-Wurttemberg
  - Universitatsklinik Regensburg /ID# 137920, Regensburg, Bavaria
  - Univ Klinik Eppendorf Hamburg /ID# 137921, Hamburg
  - LMU Klinikum der Universität München /ID# 137922, Munich
  - Universitatsklinikum Tubingen /ID# 137923, Tübingen
- Hungary (5):
  - Pecsi Tudomanyegyetem /ID# 136111, Pécs, Pecs
  - Semmelweis Egyetem /ID# 152578, Budapest
  - National Institute of Oncology /ID# 135970, Budapest
  - Orszagos Klinikai Idegtudomany /ID# 135971, Budapest
  - Debreceni Egyetem Klinikai Központ /ID# 135969, Debrecen
- Ireland (2):
  - Cork University Hospital /ID# 136828, Cork
  - Beaumont Hospital /ID# 136829, Dublin
- Italy (5):
  - Ospedale Bellaria.Azienda USL IRCCS.Istituto delle Scienze Neurologiche di Bolog /ID# 138335, Bologna
  - Ospedale Generale di Bolzano /ID# 138338, Bolzano
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 140395, Milan
  - Istituto Oncologico Veneto /ID# 138336, Padua
  - Azienda Ospedaliera Sant' Andrea /ID# 138337, Rome
- Hospital Zambrano Hellion /ID# 138076, San Pedro Garza García, Mexico
- Netherlands (6):
  - Vrije Universiteit Medisch Centrum /ID# 137221, Amsterdam
  - Universitair Medisch Centrum Groningen /ID# 138266, Groningen
  - Erasmus Medisch Centrum /ID# 136981, Rotterdam
  - Haaglanden Medisch Centrum /ID# 137222, The Hague
  - Universitair Medisch Centrum Utrecht /ID# 137219, Utrecht
  - Prinses Maxima Centrum /ID# 204409, Utrecht
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne /ID# 137919, Gdansk, Masovian Voivodeship
  - Wojewodzkie Wielospecjalistycz /ID# 137654, Lodz
- Singapore (3):
  - National University Hospital /ID# 135951, Singapore
  - National Cancer Ctr Singapore /ID# 135952, Singapore
  - KK Women's & Children Hospital /ID# 153676, Singapore
- South Korea (3):
  - Seoul National Univ Bundang ho /ID# 136841, Seongnam, Gyeonggido
  - Samsung Medical Center /ID# 136842, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 136840, Seoul
- Spain (5):
  - Instituto Catalán de Oncología (ICO) Badalona /ID# 140976, Badalona, Barcelona
  - Clinica Universitar de Navarra - Pamplona /ID# 140047, Pamplona, Navarra, Comunidad
  - Instituto Catalan de Oncologia (ICO) & Hosp. de Bellvitge /ID# 137688, Barcelona
  - Hospital Universitario Nino /ID# 153800, Madrid
  - Hosp Univ 12 de Octubre /ID# 137908, Madrid
- Switzerland (2):
  - Centre Hospitalier Univ Vaudoi /ID# 137929, Lausanne
  - University Hospital Zurich /ID# 137930, Zurich
- Taiwan (5):
  - China Medical University Hosp /ID# 136976, Taichung, Taichung
  - National Taiwan Univ Hosp /ID# 136975, Taipei City, Taipei
  - Taichung Veterans General Hosp /ID# 136977, Taichung
  - Taipei Veterans General Hosp /ID# 136974, Taipei
  - Linkou Chang Gung Memorial Ho /ID# 136944, Taoyuan
- United Kingdom (7):
  - Guy's and St Thomas' NHS Found /ID# 140312, London, London, City of
  - Univ Hospitals Birmingham NHS Foundation trust /ID# 136978, Birmingham
  - Gartnavel General Hospital /ID# 136979, Glasgow
  - Hull and East Yorkshire NHS /ID# 136917, Hull
  - University College Hospitals /ID# 136879, London
  - Great Ormond St Hospital NHS /ID# 153421, London
  - Christie NHS Foundation Trust /ID# 140313, Manchester

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Clement PMJ, Dirven L, Eoli M, Sepulveda-Sanchez JM, Walenkamp AME, Frenel JS, Franceschi E, Weller M, Chinot O, De Vos FYFL, Whenham N, Sanghera P, Looman J, Kundu MG, Peter de Geus J, Nuyens S, Spruyt M, Gorlia T, Coens C, Golfinopoulos V, Reijneveld JC, van den Bent MJ. Impact of depatuxizumab mafodotin on health-related quality of life and neurological functioning in the phase II EORTC 1410/INTELLANCE 2 trial for EGFR-amplified recurrent glioblastoma. Eur J Cancer. 2021 Apr;147:1-12. doi: 10.1016/j.ejca.2021.01.010. Epub 2021 Feb 15. PMID 33601293
- [Derived] Van Den Bent M, Eoli M, Sepulveda JM, Smits M, Walenkamp A, Frenel JS, Franceschi E, Clement PM, Chinot O, De Vos F, Whenham N, Sanghera P, Weller M, Dubbink HJ, French P, Looman J, Dey J, Krause S, Ansell P, Nuyens S, Spruyt M, Brilhante J, Coens C, Gorlia T, Golfinopoulos V. INTELLANCE 2/EORTC 1410 randomized phase II study of Depatux-M alone and with temozolomide vs temozolomide or lomustine in recurrent EGFR amplified glioblastoma. Neuro Oncol. 2020 May 15;22(5):684-693. doi: 10.1093/neuonc/noz222. PMID 31747009
- [Derived] Lassman AB, van den Bent MJ, Gan HK, Reardon DA, Kumthekar P, Butowski N, Lwin Z, Mikkelsen T, Nabors LB, Papadopoulos KP, Penas-Prado M, Simes J, Wheeler H, Walbert T, Scott AM, Gomez E, Lee HJ, Roberts-Rapp L, Xiong H, Ansell PJ, Bain E, Holen KD, Maag D, Merrell R. Safety and efficacy of depatuxizumab mafodotin + temozolomide in patients with EGFR-amplified, recurrent glioblastoma: results from an international phase I multicenter trial. Neuro Oncol. 2019 Jan 1;21(1):106-114. doi: 10.1093/neuonc/noy091. PMID 29982805
- [Derived] Gan HK, Reardon DA, Lassman AB, Merrell R, van den Bent M, Butowski N, Lwin Z, Wheeler H, Fichtel L, Scott AM, Gomez EJ, Fischer J, Mandich H, Xiong H, Lee HJ, Munasinghe WP, Roberts-Rapp LA, Ansell PJ, Holen KD, Kumthekar P. Safety, pharmacokinetics, and antitumor response of depatuxizumab mafodotin as monotherapy or in combination with temozolomide in patients with glioblastoma. Neuro Oncol. 2018 May 18;20(6):838-847. doi: 10.1093/neuonc/nox202. PMID 29077941
- [Derived] Reardon DA, Lassman AB, van den Bent M, Kumthekar P, Merrell R, Scott AM, Fichtel L, Sulman EP, Gomez E, Fischer J, Lee HJ, Munasinghe W, Xiong H, Mandich H, Roberts-Rapp L, Ansell P, Holen KD, Gan HK. Efficacy and safety results of ABT-414 in combination with radiation and temozolomide in newly diagnosed glioblastoma. Neuro Oncol. 2017 Jul 1;19(7):965-975. doi: 10.1093/neuonc/now257. PMID 28039367

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intention-to-treat population (ITT): all randomized participants. Nine enrolled adult participants did not have a screen failure form reported and were not randomized. In the table below, "Completed" and "Not completed" refer to study drug treatment, and the reasons not completed listings refer to study drug treatment.
Period: Overall Study
Arm/Group | ABT-414/Temozolomide | ABT-414_adult | Control_lomustine | Control_ Temozolomide | ABT-414_ Pediatric
Started | 88 | 86 | 60 | 26 | 6
Completed | 0 | 0 | 2 | 0 | 1
Not Completed | 88 | 86 | 58 | 26 | 5
Not completed — Progressive disease | 72 | 70 | 43 | 15 | 5
Not completed — Adverse Event | 6 | 8 | 6 | 3 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 8 | 3 | 0
Not completed — Death | 2 | 1 | 0 | 0 | 0
Not completed — Start of a new anti-cancer treatment | 0 | 1 | 0 | 1 | 0
Not completed — Other primary malignancy | 0 | 1 | 0 | 0 | 0
Not completed — Other, not specified | 2 | 1 | 1 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population (ITT): all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | ABT-414/Temozolomide | ABT-414_adult | Control_lomustine | Control_ Temozolomide | ABT-414_ Pediatric | Total
Number analyzed (Participants) | 88 | 86 | 60 | 26 | 6 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (8.15) | 58.1 (9.18) | 57.8 (10.62) | 55.9 (11.04) | 10.5 (5.43) | 56.7 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 36 | 19 | 9 | 5 | 98
  Male | 59 | 50 | 41 | 17 | 1 | 168
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 7 | 5 | 2 | 0 | 22
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  White | 16 | 6 | 12 | 4 | 3 | 41
  Other | 0 | 0 | 0 | 0 | 0 | 0
  Not Reported | 0 | 0 | 0 | 1 | 0 | 1
  Missing | 64 | 73 | 43 | 19 | 3 | 202

OUTCOME MEASURES:

1. Primary Outcome: Adult Study: Overall Survival (OS)
Description: Overall Survival (OS) was defined as time from randomization to death due to any cause, regardless of whether the event occurred on or off study drug (depatuxizumab mafodotin/temozolomide/lomustine).
Time Frame: From the date of randomization up to the date of participant's death; participants who completed treatment were to be assessed every 12 weeks, up to 28 months.
Population: All randomized adult participants; participants in the control arms were treated based on the time of relapse and they differ in prognostic profile, therefore data were combined.
Measure: Number (95% Confidence Interval); unit: months
Groups:
- Control (Temozolomide/Lomustine): Adult participants relapsing during temozolomide (TMZ) treatment or within the first 16 weeks after the first day of the last TMZ cycle who received lomustine on Day 1 of every 42-day treatment period until one of the treatment withdrawal criteria was met, up to a maximum of 1 year OR adult subjects relapsing 16 weeks or more after the first day of the last temozolomide (TMZ) cycle who received TMZ on Day 1 to Day 5 for the first 28-day cycle, with dose escalation in subsequent cycles in case of adequate tolerance and treatment continuing until one of the treatment withdrawal criteria was met.
Arm/Group | ABT-414/Temozolomide | ABT-414_adult | Control (Temozolomide/Lomustine)
Number analyzed (Participants) | 88 | 86 | 86
months
  25th quartile | 5.7 [4.0 to 6.8] | 4.6 [3.5 to 5.5] | 4.9 [4.1 to 5.4]
  50th quartile | 9.6 [7.4 to 11.8] | 7.9 [6.1 to 8.7] | 8.2 [5.9 to 9.5]
  75th quartile | 16.9 [14.4 to NA] — Not calculable due to insufficient number of participants with events | 15.5 [10.2 to 19.0] | 12.6 [10.2 to 14.9]
Statistical Analysis 1: Comparison: ABT-414/Temozolomide vs Control (Temozolomide/Lomustine); Stratified at randomization by regions of the world (North America, Europe and Australia, Asia/Other Regions), WHO performance status (0, > 0), timing of relapse (< 16 weeks, ≥ 16 weeks after first day of last TMZ cycle); Test type: Other; p = 0.062, Log Rank — 2-sided; Cox Proportional Hazard = 0.71, 95% CI 2-sided [0.5 to 1.02]
Statistical Analysis 2: Comparison: ABT-414_adult vs Control (Temozolomide/Lomustine); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.835, Log Rank — 2-sided; Cox Proportional Hazard = 1.04, 95% CI 2-sided [0.73 to 1.48]

2. Primary Outcome: Adult Study: Progression-Free Survival (PFS)
Description: Progression-free survival was assessed per response assessment in neuro-oncology criteria (RANO) criteria and assessed by an independent review committee and was defined as the length of time during and after the treatment of a disease, that the participant lived with the disease but did not get worse.
Time Frame: Measured every 8 weeks from date of randomization until the date of first objective progression or subject's death, whichever occurred first, up to 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | ABT-414/Temozolomide | ABT-414_adult | Control (Temozolomide/Lomustine)
Number analyzed (Participants) | 88 | 86 | 86
months
  25th quartile | 1.8 [1.7 to 2.0] | 1.5 [1.1 to 1.7] | 1.6 [1.3 to 1.7]
  50th quartile | 2.7 [2.0 to 3.8] | 1.9 [1.8 to 2.0] | 1.9 [1.9 to 2.2]
  75th quartile | 4.9 [3.9 to 9.3] | 3.5 [2.1 to 3.9] | 4.2 [3.4 to 5.8]
Statistical Analysis 1: Comparison: ABT-414/Temozolomide vs Control (Temozolomide/Lomustine); Test type: Other; p = 0.123, Log Rank — 2-sided; Cox Proportional Hazard = 0.77, 95% CI 2-sided [0.55 to 1.07]
Statistical Analysis 2: Comparison: ABT-414_adult vs Control (Temozolomide/Lomustine); Test type: Other; p = 0.117, Log Rank — 2-sided; Cox Proportional Hazard = 1.31, 95% CI 2-sided [0.93 to 1.84]

3. Primary Outcome: Pediatric Study: Percentage of Participants With Adverse Events From the First Visit Until 49 Days After the Last Dose of Study Drug
Description: The severity of each adverse event was rated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE Version 4.0)
Time Frame: From participant's first visit until 49 days after the participant's last dose of study drug, up to 63 weeks
Population: Pediatric participants (safety population)
Measure: Number; unit: percentage of participants
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 6
percentage of participants | 100

4. Primary Outcome: Pediatric Study: Maximum Observed Serum Concentration (Cmax) of ABT-414
Description: Cmax is the peak concentration that a drug achieves in a specified compartment after the drug has been administrated and before administration of a second dose.
Time Frame: Samples collected Cycle 1 Days 1, 2,3,5,8,15; Cycle 2 Day 1; Cycle 3 Day 1; Cycle 5 Day 1; Day 1 of every two cycles starting with Cycle 5; and 35 days after the last dose
Population: Pediatric participants with available data
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 5
µg/mL | 31.4 (15.0)

5. Primary Outcome: Pediatric Study: Maximum Observed Plasma Concentration (Cmax) of Cys-mcMMAF
Description: Cmax is the peak concentration that a drug or drug metabolite achieves in a specified compartment after the drug has been administrated and before administration of a second dose. Cys-mcMMAF is a toxic metabolite of depatuxizumab mafodotin.
Time Frame: Samples collected Cycle 1 Days 1, 2, 3, 5, 8
Population: Pediatric participants with available data
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 5
ng/mL | 0.272 (0.0983)

6. Primary Outcome: Pediatric Study: Half-life (t1/2) Observed for ABT-414
Description: Half-life is the calculated time it takes for half of the drug to leave the body.
Time Frame: as for outcome 4
Population: Pediatric participants with available data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 4
days | 9.0 (1.5)

7. Primary Outcome: Pediatric Study: Half-life (t1/2) Observed for Cys-mcMMAF
Description: Half-life is the calculated time it takes for half of the drug or drug metabolite to leave the body. CysmcMMAF is a toxic metabolite of depatuxizumab mafodotin.
Time Frame: Samples collected Cycle 1 Days 1, 2, 3, 5, 8
Population: Pediatric participants with available data
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 2
days | 11.2 (22.9)

8. Primary Outcome: Pediatric Study: Area Under the Concentration-time Curve (AUC) Observed for ABT-414
Description: AUC is a measure of how long and how much drug is present in the body after dosing. The AUC of depatuxizumab mafodotin (ABT-414) in the pediatric population was measured following treatment to confirm that this was comparable to adults, and that the dosing levels are appropriate for a pediatric population.
Time Frame: as for outcome 4
Population: Pediatric participants with available data
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 5
µg*h/mL | 3170 (1320)

9. Primary Outcome: Pediatric Study: Area Under the Concentration-time-curve (AUC) Observed for Unconjugated Cys-mcMMAF
Description: AUC is a measure of how long and how much drug or drug metabolite is present in the body after dosing. The AUC of Cys-mcMMAF, a toxic metabolite of depatuxizumab mafodotin, in the pediatric population was measured following treatment to confirm that this was comparable to adults, and that the dosing levels are appropriate for a pediatric population.
Time Frame: Samples collected Cycle 1 Days 1, 2, 3, 5, 8
Population: Pediatric participants with available data
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 5
ng*h/mL | 14.1 (6.22)

10. Secondary Outcome: Adult Study: Objective Response Rate (ORR)
Description: The objective response rate (ORR) included best overall responses - complete response (CR) and partial response (PR) - assessed by the independent review committee per response assessment in neurooncology criteria (RANO) criteria from the date of randomization until disease progression or death, whichever came first. All objective responses (CR and PR) must be have been confirmed by repeat MRI 4 weeks after the first time when CR or PR is identified. Any subject who did not meet CR or PR including those who did not have post-baseline radiological assessments was considered a nonresponder.
Time Frame: Every 8 weeks at each assessment of disease, up to 28 months
Population: Participants with measurable disease at baseline; participants in the control arms were treated based on the time of relapse and they differ in prognostic profile, therefore data were combined.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABT-414/Temozolomide | ABT-414_adult | Control (Temozolomide/Lomustine)
Number analyzed (Participants) | 49 | 39 | 45
percentage of participants | 14.3 [5.9 to 27.2] | 7.7 [1.6 to 20.9] | 4.4 [0.5 to 15.1]
Statistical Analysis 1: Comparison: ABT-414/Temozolomide vs Control (Temozolomide/Lomustine); Comparison is based on Cochran-Mantel-Haenszel method with stratification factors. Stratified at randomization by regions of the world (North America, Europe and Australia, Asia/Other Regions), WHO performance status (0, > 0), timing of relapse (< 16 weeks, ≥ 16 weeks after first day of last TMZ cycle); Test type: Other; p = 0.06, Cochran-Mantel-Haenszel — 2-sided; Odds Ratio (OR) = 3.1, 95% CI 2-sided [0.6 to 16.16]
Statistical Analysis 2: Comparison: ABT-414_adult vs Control (Temozolomide/Lomustine); [analysis description as in outcome 10, analysis 1]; Test type: Other; p = 0.767, Cochran-Mantel-Haenszel — 2-sided; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.12 to 12.49]

11. Secondary Outcome: Adult Study: Overall Survival in the Subgroup With Epidermal Growth Factor Receptor (EGFRvIII) Mutation
Description: Overall Survival (OS) was defined as time from randomization to death due to any cause, regardless of whether the event occurred on or off study drug (depatuxizumab mafodotin/temozolomide/lomustine) for all randomized participants that had the Epidermal Growth Factor Receptor (EGFRvIII) mutation.
Time Frame: as for outcome 1
Population: Randomized adult participants with EGFRvIII-mutated tumors; participants in the control arms were treated based on the time of relapse and they differ in prognostic profile, therefore data were combined.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | ABT-414/Temozolomide | ABT-414_adult | Control (Temozolomide/Lomustine)
Number analyzed (Participants) | 39 | 36 | 47
months
  25th quartile | 6.3 [3.1 to 7.4] | 5.0 [3.1 to 5.9] | 4.7 [3.0 to 5.8]
  50th quartile | 9.4 [7.1 to 11.0] | 8.4 [5.5 to 9.0] | 7.5 [5.1 to 9.6]
  75th quartile | 14.4 [10.3 to NA] — Not calculable due to insufficient number of participants with events | 13.9 [8.7 to NA] — Not calculable due to insufficient number of participants with events | 12.4 [9.5 to 16.2]
Statistical Analysis 1: Comparison: ABT-414/Temozolomide vs Control (Temozolomide/Lomustine); Test type: Other; p = 0.127, Log Rank — 2-sided; Cox Proportional Hazard = 0.67, 95% CI 2-sided [0.4 to 1.13]
Statistical Analysis 2: Comparison: ABT-414_adult vs Control (Temozolomide/Lomustine); Test type: Other; p = 0.64, Log Rank — 2-sided; Cox Proportional Hazard = 0.88, 95% CI 2-sided [0.52 to 1.49]

12. Secondary Outcome: Pediatric Study: Objective Response Rate (ORR)
Description: The pediatric data collection for this study was still ongoing when INTELLANCE-1 (NCT02573324; EudraCT number 2015-001166-26) interim efficacy results overall indicated no survival benefit to adding depatuxizumab mafodotin to standard radiotherapy/temozolomide therapy in newly diagnosed glioblastoma patients. Based on the INTELLANCE-1 results, AbbVie decided to stop further enrollment of pediatric participants into the pediatric substudy and to stop the collection of efficacy data. Because of this decision not to summarize except for safety data, the pediatric substudy ORR analysis was not summarized due to the small number of pediatric participants enrolled in the study.
Time Frame: Evaluated every 8 weeks (+/- 7 days) at each assessment of disease according to response assessment in neuro-oncology criteria (RANO), until progression or withdrawal up to approximately 52 weeks
Population: Pediatric efficacy data were not collected
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 0

13. Secondary Outcome: Pediatric Study: Best Tumor Response Rate
Description: as for outcome 12
Time Frame: as for outcome 12
Population: Pediatric efficacy data were not collected
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 0

14. Secondary Outcome: Pediatric Study: Duration of Response
Description: as for outcome 12
Time Frame: as for outcome 12
Population: Pediatric efficacy data were not collected
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 0

15. Secondary Outcome: Pediatric Study: Overall Survival
Description: as for outcome 12
Time Frame: From the date of enrollment to the date of death; participants who completed treatment were to be assessed every 12 weeks, up to 28 months
Population: Pediatric efficacy data were not collected
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 0

16. Secondary Outcome: Pediatric Study: Time to Progression
Description: The pediatric data collection for this study was still ongoing when INTELLANCE-1 (NCT02573324; EudraCT number 2015-001166-26) interim efficacy results overall indicated no survival benefit to adding depatuxizumab mafodotin to standard radiotherapy/ temozolomide therapy in newly diagnosed glioblastoma patients. Based on the INTELLANCE-1 results, AbbVie decided to stop further enrollment of pediatric participants into the pediatric substudy and to stop the collection of efficacy data. Because of this decision not to summarize except for safety data, pediatric time to progression data analysis was not summarized due to the small number of pediatric participants enrolled in the study.
Time Frame: Evaluated every 8 weeks (+/- 7 days) from the date of enrollment until the date of first objective progression or participant's death, whichever occurs first, up to approximately 52 weeks
Population: Pediatric efficacy data were not collected
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 0

17. Secondary Outcome: Pediatric Study: Progression-Free Survival
Description: as for outcome 12
Time Frame: as for outcome 16
Population: Pediatric efficacy data were not collected
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 0

18. Secondary Outcome: Pediatric Study: Percentage of Participants With Changes in Neurological Status and Functioning
Description: as for outcome 12
Time Frame: Baseline, Day 1 and 15 of each cycle, every 6 months for 5 years thereafter, and then annually
Population: Pediatric efficacy data were not collected
Arm/Group | ABT-414_ Pediatric
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 35 days (adults) or 49 days (pediatric subjects) after the last dose of study drug, up to 125 weeks.
Description: Serious and non-serious adverse events occurring after the subject signed the study-specific informed consent and prior to the initial dose of study drug were to be collected only if they were considered by the Investigator to be causally related to required study procedures.
Groups:
- ABT-414/Temozolomide: Depatuxizumab mafodotin (ABT-414) administered once every 2 weeks in combination with temozolomide (TMZ) to adult subjects
- ABT-414_adult: Depatuxizumab mafodotin (ABT-414) administered once every 2 weeks to adult subjects
- Control_lomustine: Adult subjects relapsing during temozolomide (TMZ) treatment or within the first 16 weeks after the first day of the last TMZ cycle received lomustine on Day 1 of every 42-day treatment period until one of the treatment withdrawal criteria was met, up to a maximum of 1 year.
- Control_ Temozolomide: Adult subjects relapsing 16 weeks or more after the first day of the last temozolomide (TMZ) cycle received TMZ on Day 1 to Day 5 for the first 28-day cycle, with dose escalation in subsequent cycles in case of adequate tolerance and treatment continuing until one of the treatment withdrawal criteria was met.
Arm/Group | ABT-414/Temozolomide | ABT-414_adult | Control_lomustine | Control_ Temozolomide | ABT-414_ Pediatric
All-Cause Mortality (participants affected / at risk) | 80/88 | 80/84 | 52/56 | 21/21 | 5/6
Serious Adverse Events (participants affected / at risk) | 39/88 | 30/84 | 19/56 | 5/21 | 3/6
Other Adverse Events (participants affected / at risk) | 84/88 | 76/84 | 46/56 | 20/21 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-414/Temozolomide (N=88) | ABT-414_adult (N=84) | Control_lomustine (N=56) | Control_ Temozolomide (N=21) | ABT-414_ Pediatric (N=6)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CORNEAL EPITHELIAL MICROCYSTS (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (4)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENINGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (16) | 7 (10) | 2 (4) | 2 (2) | 2 (2)
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APRAXIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPILEPSY (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEMIPLEGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASTICITY (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
NEUROLOGICAL DECOMPENSATION (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
PARTIAL SEIZURES (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 9 (9) | 3 (3) | 4 (4) | 1 (1) | 0 (0)
STATUS EPILEPTICUS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBDURAL HYGROMA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBGALEAL HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-414/Temozolomide (N=88) | ABT-414_adult (N=84) | Control_lomustine (N=56) | Control_ Temozolomide (N=21) | ABT-414_ Pediatric (N=6)
ANAEMIA (Blood and lymphatic system disorders) | 7 (7) | 4 (13) | 5 (7) | 0 (0) | 1 (1)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 5 (11) | 1 (4) | 0 (0)
LYMPHOPENIA (Blood and lymphatic system disorders) | 9 (17) | 8 (16) | 9 (13) | 4 (8) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 1 (3) | 10 (12) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 19 (55) | 7 (11) | 19 (34) | 8 (11) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
CUSHINGOID (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CATARACT (Eye disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
CORNEAL EPITHELIAL MICROCYSTS (Eye disorders) | 25 (64) | 12 (22) | 0 (0) | 0 (0) | 1 (1)
CORNEAL OPACITY (Eye disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 20 (36) | 22 (33) | 1 (1) | 0 (0) | 2 (2)
EYE IRRITATION (Eye disorders) | 6 (8) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
EYE PAIN (Eye disorders) | 7 (10) | 11 (20) | 0 (0) | 0 (0) | 2 (2)
EYELID PTOSIS (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
KERATITIS (Eye disorders) | 16 (24) | 27 (45) | 0 (0) | 0 (0) | 1 (1)
KERATOPATHY (Eye disorders) | 15 (24) | 7 (8) | 0 (0) | 0 (0) | 3 (3)
LACRIMATION INCREASED (Eye disorders) | 9 (10) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
OCULAR DISCOMFORT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHOTOPHOBIA (Eye disorders) | 12 (14) | 8 (11) | 0 (0) | 0 (0) | 3 (4)
PUNCTATE KERATITIS (Eye disorders) | 3 (6) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
PUPILLARY REFLEX IMPAIRED (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 30 (52) | 17 (27) | 1 (1) | 0 (0) | 2 (5)
VISUAL IMPAIRMENT (Eye disorders) | 3 (3) | 5 (6) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 23 (28) | 8 (9) | 2 (2) | 6 (6) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 8 (9) | 6 (6) | 3 (3) | 1 (1) | 1 (2)
NAUSEA (Gastrointestinal disorders) | 21 (33) | 8 (8) | 6 (6) | 6 (7) | 2 (3)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 19 (23) | 5 (5) | 3 (4) | 6 (6) | 3 (5)
ASTHENIA (General disorders) | 6 (9) | 3 (4) | 4 (7) | 2 (2) | 1 (1)
FATIGUE (General disorders) | 33 (60) | 27 (39) | 13 (16) | 5 (6) | 2 (6)
GAIT DISTURBANCE (General disorders) | 4 (5) | 3 (5) | 2 (2) | 2 (2) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 7 (9) | 2 (2) | 4 (5) | 4 (4) | 0 (0)
PYREXIA (General disorders) | 5 (5) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
CONJUNCTIVITIS (Infections and infestations) | 7 (8) | 6 (6) | 1 (1) | 0 (0) | 1 (1)
EYE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 5 (6) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VAGINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 4 (5) | 4 (5) | 3 (3) | 0 (0) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 11 (24) | 12 (17) | 3 (4) | 1 (1) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 9 (12) | 13 (15) | 2 (2) | 0 (0) | 1 (4)
BLOOD CULTURE POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 4 (6) | 8 (15) | 0 (0) | 0 (0) | 0 (0)
LYMPHOCYTE COUNT DECREASED (Investigations) | 7 (11) | 4 (4) | 6 (13) | 2 (2) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1) | 8 (11) | 1 (1) | 1 (10)
PLATELET COUNT DECREASED (Investigations) | 21 (46) | 9 (17) | 15 (31) | 2 (6) | 1 (29)
WEIGHT DECREASED (Investigations) | 4 (4) | 7 (9) | 3 (4) | 0 (0) | 3 (8)
WEIGHT INCREASED (Investigations) | 6 (8) | 6 (9) | 3 (3) | 1 (1) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 (7) | 2 (2) | 5 (15) | 1 (1) | 2 (8)
DECREASED APPETITE (Metabolism and nutrition disorders) | 10 (11) | 5 (7) | 2 (2) | 0 (0) | 1 (2)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 5 (8) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 7 (12) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (8) | 7 (7) | 4 (4) | 2 (2) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
APHASIA (Nervous system disorders) | 9 (10) | 9 (10) | 3 (3) | 3 (3) | 0 (0)
ATAXIA (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
BALANCE DISORDER (Nervous system disorders) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 7 (9) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 3 (3) | 3 (4) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 21 (31) | 20 (21) | 8 (8) | 2 (2) | 2 (3)
HEMIPARESIS (Nervous system disorders) | 2 (2) | 7 (7) | 7 (9) | 0 (0) | 2 (2)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 6 (13) | 7 (11) | 5 (9) | 1 (1) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 3 (3) | 3 (3) | 3 (6) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 5 (6) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
DEPRESSION (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
DISINHIBITION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 8 (10) | 6 (7) | 2 (2) | 2 (2) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 2 (2) | 3 (3) | 3 (3) | 2 (2)
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 1 (1)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (3) | 1 (1) | 2 (2) | 0 (0)
HYPERTENSION (Vascular disorders) | 9 (18) | 6 (9) | 4 (5) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-01-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT02343406/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT02343406/SAP_001.pdf